CLINICAL TRIAL: NCT03905707
Title: A Double-Blind Phase 3 Extension Trial Assessing the Long Term Safety and Efficacy of Glepaglutide in Patients With Short Bowel Syndrome (SBS)
Brief Title: Evaluation of Long Term Safety and Efficacy of Glepaglutide in Treatment of SBS
Acronym: EASE SBS 2
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP1848-17127
Record Dates: First submitted 2019-03-28; First posted 2019-04-05 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Short Bowel Syndrome
MeSH Terms: conditions — Short Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glepaglutide SC injections twice weekly (Experimental): Glucagon-Like Peptide-2 (GLP-2) analog, 10 mg subcutaneous injection twice weekly.
  In this long term safety study, there is no placebo arm.
  Interventions: Drug: glepaglutide
- Glepaglutide SC injections once weekly and placebo once weekly (Experimental): Glucagon-Like Peptide-2 (GLP-2) analog, 10 mg subcutaneous injection once weekly and placebo once weekly.
  In this long term safety study, there is no placebo arm.
  Interventions: Drug: glepaglutide

INTERVENTIONS:
Drug: glepaglutide — Glucagon-Like Peptide-2 (GLP-2) analog
  Other Names: ZP1848

SUMMARY:
The primary objective of the trial is to evaluate the long-term safety of glepaglutide treatment in patients with short bowel syndrome (SBS).

Glepaglutide is the International Nonproprietary Name and USAN for ZP1848.

DETAILED DESCRIPTION:
A Double-Blind Phase 3 Extension Trial Assessing the Long Term Safety and Efficacy of Glepaglutide in Patients with Short Bowel Syndrome (SBS)

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activity
* Completed the lead-in trial (ZP1848-17111) or completed the Phase 2 trial (ZP1848-15073)

Exclusion Criteria:

* Withdrawal of consent from the lead-in trial
* Any condition or disease or circumstance that in the Investigator's opinion would put the patient at any undue risk, prevent completion of the trial, or interfere with the analysis of the trial results
* Use of GLP-1, GLP-2, human growth hormone, somatostatin, or analogs thereof, within 3 months prior to Screening
* Females of childbearing potential, who are pregnant, breast-feeding, intend to become pregnant or are not using highly effective contraceptive methods

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2019-05-07 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse Events | 2 years
  Incidence and type of Adverse Events

SECONDARY OUTCOMES:
Safety - Serious Adverse Events | 2 years
  Incidence and type of Serious Adverse Events
Safety - Adverse Events of Special Interest | 2 years
  Incidence and type of Adverse Events of Special Interest
Safety - Changes in blood pressure from baseline | 2 years
  Changes in systolic and diastolic blood pressure will be reported
Number of patients with clinically significant changes in 12-Lead electrocardiogram (ECG) | 2 years
  Number of patients with clinically significant changes in ECG will be reported
Immunogenicity - Occurrence of anti-drug antibodies | 2 years
  Occurrence of antibodies against glepaglutide
Change in weekly Parenteral Support (PS) volume | 2 years
  Change in weekly PS volume from baseline
Number of patients with 20 percent reduction in PS volume | 2 years
  Achieving at least 20 percent reduction in weekly PS volume from baseline
Days off PS | 2 years
  Achieving 1 or more days per week off PS
Weaned off PS | 2 years
  Reduction in weekly PS volume of 100 percent (weaned off)
Changes in fluid composite effect | 2 years
  Reduction in PS plus reduction in oral fluid intake plus increase in urine volume from baseline
Energy content (lipids) | 2 years
  Change in lipids content (in kcal/L or kjoule/L) of PS from baseline
Energy content (glucose) | 2 years
  Change in glucose content (in kcal/L or kjoule/L) of PS from baseline
Energy content (amino acids) | 2 years
  Change in amino acids content (in kcal/L or kjoule/L) of PS from baseline
Days on PS | 2 years
  Change in number of days on PS per week from baseline
Number of patients with 40 percent change in PS volume per week | 2 years
  Achieving 40 percent in PS volume from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Zealand Pharma, Study Director — Zealand Pharma
Locations (27):
- United States (7):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Children's Hospital, Chicago, Illinois
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Nashville, Tennessee
- UZ Leuven, Leuven, Belgium
- Canada (3):
  - The Royal Alexandra Hospital, Edmonton
  - Western University, London
  - University Health Network - Toronto General Hospital, Toronto
- Rigshospitalet, Copenhagen, Denmark
- France (2):
  - Hôpital Beaujon, Clichy
  - Centre Hospitalier Lyon-Sud, Pierre-Bénite
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Bonn, Bonn
  - Universitätsklinikum Frankfurt - Med. Klinik I, Frankfurt
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Universitätsmedizin Rostock, Rostock
- UMC Radboud Nijmegen, Nijmegen, Netherlands
- Poland (3):
  - Wojewodzki Specjalistyczny Szpital im. M. Pirogowa w Lodzi, Lodz
  - Solumed, Poznan
  - Szpital Skawina sp. z o.o. im. Stanley Dudricka, Skawina
- United Kingdom (4):
  - St Mark's Hospital, Harrow
  - UCLH Foundation NHS Trust, London
  - University of East Anglia, Norwich
  - University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: Undecided